CLINICAL TRIAL: NCT07015242
Title: The CAROLYN Trial: Lisocabtagene Maraleucelas First-Line Therapy for Primary Central Nervous System Lymphoma (PCNSL) in Transplant-Ineligible Patients
Brief Title: A Study of the Efficacy and Safety of Lisocabtagene Maraleucel (Liso-cel) as First-Line Therapy in Adults With Transplant-Ineligible Primary Central Nervous System Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA082-1215; 2025-521144-38 (Other: EU CTR); U1111-1318-3732 (Other: WHO)
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Rituximab; Methotrexate; Procarbazine; Temozolomide; fludarabine; Cyclophosphamide; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Liso-cel Administration (Experimental)
  Interventions: Drug: Rituximab; Drug: Methotrexate; Drug: Procarbazine; Drug: Temozolomide; Biological: Liso-cel; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Calcium folinate

INTERVENTIONS:
Drug: Rituximab — Specified dose on specified days
Drug: Methotrexate — Specified dose on specified days
Drug: Procarbazine — Specified dose on specified days
Drug: Temozolomide — Specified dose on specified days
Biological: Liso-cel — Specified dose on specified days
  Other Names: JCAR017; Breyanzi
Drug: Fludarabine — Specified dose on specified days
Drug: Cyclophosphamide — Specified dose on specified days
Drug: Calcium folinate — Specified dose on specified days
  Other Names: Leucovorin

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of lisocabtagene maraleucel (Breyanzi/liso-cel/BMS-986387) in adults as first-line treatment in transplant-ineligible Primary Central Nervous System Lymphoma (PCNSL).

ELIGIBILITY:
Inclusion Criteria

* Participant must be 18 years or older at the time of signing the informed consent form (ICF).
* Histologically confirmed primary central nervous system (CNS) lymphoma (PCNSL) prior to screening, as assessed by local pathology.
* Transplant-ineligible based on physician's assessment and meeting at least one of the following criteria: age ≥65 years or HCT-CI (Hematopoietic Cell Transplantation-specific Comorbidity Index) score ≥3.
* Participant must be suitable, per investigator, to receive a high dose methotrexate (HD-MTX) based treatment regimen.
* Prior to signing ICF, anti-cancer therapy for the treatment of PCNSL must only include standard of care regimens, with or without corticosteroids given for disease-related symptoms.
* Prior to ICF signature, participant's disease must be sensitive to prior high-dose methotrexate-based regimens, as demonstrated by a complete response (CR, no remaining signs of PCNSL) or a partial response (PR, signs of PNCSL mostly gone) per Investigator's assessment, based on the International Primary CNS Lymphoma Collaborative Group (IPCG) criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Individuals of childbearing potential (IOCBP) must have a negative highly sensitive pregnancy test within 24 hours prior to the start of study intervention.

Exclusion Criteria

* Participant has a diagnosis of secondary CNS lymphoma due to systemic disease.
* Primary intraocular lymphoma (PIOL)/ Primary vitreoretinal lymphoma (PVRL) and isolated cerebrospinal fluid (CSF) disease.
* Any significant medical condition including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she was to participate in the study based on investigator's judgement.
* History of another primary malignancy that has not been in remission for ≥2 years.
* Prior treatment with CAR T-cell or any other gene therapy product that utilizes human genome-editing technology.
* History of or active human immunodeficiency virus (HIV).
* Active hepatitis B or active hepatitis C.
* Active autoimmune disease requiring immunosuppressive therapy.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2028-01-09 (Estimated); Study Completion 2028-12-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | 12 months after liso-cel infusion
  Defined as the time from the date of liso-cel infusion to the date of first documented disease relapse or progression as assessed by the investigator, or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
PFS | 12 months after date of enrollment
  Defined as the time from the date of enrollment to the date of first documented disease relapse or progression as assessed by the investigator, or death from any cause, whichever occurs first
Modified Progression-free Survival (mPFS) | 12 months after date of enrollment
  Defined as the time from the date of enrollment to the date of first documented disease relapse or progression as assessed by the investigator, or death from any cause, whichever occurs first. Disease relapse or progression prior to liso-cel infusion is considered as an event only if the patient does not achieve complete response (CR) after liso-cel infusion.
Complete Response Rate (CRR) | Up to end of study (approximately 2 years)
  Defined as proportion of patients achieving CR at any time between liso-cel infusion and the date of first documented disease relapse or progression as assessed by the investigator, initiation of a new antineoplastic therapy to treat Primary Central Nervous System Lymphoma (PCNSL), or end of study, whichever occurs first
Overall Response Rate (ORR) | Up to end of study (approximately 2 years)
  Defined as proportion of patients achieving CR or Partial Response (PR) at any time between liso-cel infusion and the date of first documented disease relapse or progression as assessed by the investigator, initiation of a new antineoplastic therapy to treat PCNSL, or end of study, whichever occurs first
Duration of Response (DoR) | 12 months after liso-cel infusion
  Defined as the time from the date of first documented disease response (complete response [CR] or partial response [PR]) achieved after liso-cel infusion to the date of first subsequent documented disease relapse or progression as assessed by the investigator, or death from any cause
Event-free Survival (EFS) | 12 months after date of enrollment
  Defined as the time from the date of enrollment to the date of first documented disease relapse or progression as assessed by the investigator, or initiation of new antineoplastic therapy to treat PCNSL, or death from any cause, whichever occurs first
Overall Survival (OS) | 12 months after date of enrollment
  Defined as the time from the date of enrollment to the date of death from any cause
Health-related quality of life (HRQoL) | Up to end of study (approximately 2 years)
  As assessed by the European Organisation for Research and Treatment of Cancer--Quality of Life C30 Questionnaire (EORTC-QLQ-30)
Health-related quality of life (HRQoL) | Up to end of study (approximately 2 years)
  As assessed by the European Organisation for Research and Treatment of Cancer--Quality of Life BN20 Questionnaire (EORTC-QLQ-BN20)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (82):
- United States (30):
  - Local Institution - 307, Stanford, California
  - Local Institution - 0305, Aurora, Colorado
  - Local Institution - 305, Aurora, Colorado
  - Local Institution - 308, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Local Institution - 0311, Chicago, Illinois
  - Local Institution - 311, Chicago, Illinois
  - Local Institution - 314, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Local Institution - 313, Boston, Massachusetts
  - Local Institution - 0316, St Louis, Missouri
  - Local Institution - 316, St Louis, Missouri
  - Local Institution - 0315, New Brunswick, New Jersey
  - Local Institution - 315, New Brunswick, New Jersey
  - Local Institution - 310, Buffalo, New York
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Local Institution - 301, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Local Institution - 302, Cleveland, Ohio
  - Local Institution - 0309, Columbus, Ohio
  - Local Institution - 309, Columbus, Ohio
  - Local Institution - 0304, Philadelphia, Pennsylvania
  - Local Institution - 304, Philadelphia, Pennsylvania
  - Local Institution - 312, Nashville, Tennessee
  - Sarah Cannon Research Institute Oncology Partners, Nashville, Tennessee
  - Local Institution - 0303, Houston, Texas
  - Local Institution - 303, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Local Institution - 306, Seattle, Washington
- France (32):
  - Local Institution - 0111, Nice, Alpes-Maritimes
  - Local Institution - 111, Nice, Alpes-Maritimes
  - Local Institution - 0104, Nantes, Loire-Atlantique
  - Local Institution - 104, Nantes, Loire-Atlantique
  - Local Institution - 0103, Pierre-Bénite, Rhône
  - Local Institution - 0106, Dijon
  - Local Institution - 106, Dijon
  - Local Institution - 0113, Lille
  - Local Institution - 113, Lille
  - Local Institution - 0112, Marseille
  - Local Institution - 112, Marseille
  - Local Institution - 0107, Montpellier
  - Local Institution - 107, Montpellier
  - Local Institution - 0114, Paris
  - Local Institution - 114, Paris
  - Local Institution - 0102, Paris
  - Local Institution - 102, Paris
  - Local Institution - 0108, Pessac
  - Local Institution - 108, Pessac
  - Local Institution - 103, Pierre-Bénite
  - CHU de Rennes - Hopital de Pontchaillou, Rennes
  - Local Institution - 101, Rennes
  - Local Institution - 0105, Rouen
  - Local Institution - 105, Rouen
  - Local Institution - 0110, Saint-Cloud
  - Local Institution - 110, Saint-Cloud
  - Local Institution - 0115, Strasbourg
  - Local Institution - 115, Strasbourg
  - Local Institution - 0109, Toulouse
  - Local Institution - 109, Toulouse
  - Local Institution - 0116, Vandœuvre-lès-Nancy
  - Local Institution - 116, Vandœuvre-lès-Nancy
- Germany (20):
  - Local Institution - 0202, Freiburg im Breisgau, Baden-Wurttemberg
  - Local Institution - 0205, Ulm, Baden-Wurttemberg
  - Local Institution - 205, Ulm, Baden-Wurttemberg
  - Local Institution - 0204, Cologne, North Rhine-Westphalia
  - Local Institution - 204, Cologne, North Rhine-Westphalia
  - Local Institution - 0206, Essen, North Rhine-Westphalia
  - Local Institution - 206, Essen, North Rhine-Westphalia
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Local Institution - 208, Chemnitz, Saxony
  - Local Institution - 0203, Berlin
  - Local Institution - 203, Berlin
  - Local Institution - 202, Freiburg im Breisgau
  - Local Institution - 0207, Göttingen
  - Local Institution - 207, Göttingen
  - Local Institution - 209, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Local Institution - 210, Heidelberg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Local Institution - 0201, Stuttgart
  - Local Institution - 201, Stuttgart

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07015242.html